CLINICAL TRIAL: NCT02588456
Title: Pilot Study of Autologous Anti-CD22 Chimeric Antigen Receptor Redirected T Cells In Patients With Chemotherapy Resistant Or Refractory Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated due to lack of efficacy
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 31415, 822967
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2018-01

CONDITIONS: Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Recurrence; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Biological: CART22 cells

INTERVENTIONS:
Biological: CART22 cells — CART22 cells transduced with a lentiviral vector to express anti-CD22 scFv TCRz:41BB administered by IV infusion.

SUMMARY:
This is a single center, single arm, open-label pilot study to determine the feasibility and safety of a single dose of autologous T cells expressing CD22 chimeric antigen receptors expressing tandem TCRζ and 4-1BB (TCRζ/4-1BB) co-stimulatory domains (referred to as "CART22" cells) administered in split fractions, in adult patients with relapsed or refractory B-cell acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form must be obtained prior to any research procedure.
2. Relapsed or refractory B-cell ALL:

   a. 1st or greater BM relapse OR b. Any marrow relapse after allogeneic HSCT and > 100 days from transplant OR c. For patients with refractory disease: i. < 60 years old that have not achieved a CR after > 2 or more chemotherapy regimens ii. >60 years old that have not achieved a CR after 1 prior chemotherapy regimen d. Patients with Ph+ ALL are eligible if they are intolerant to or have failed tyrosine kinase inhibitor therapy.

   e. Patients with CNS3 disease will be eligible if CNS disease is responsive to therapy.
3. Documentation of CD22 expression on malignant cells at relapse.
4. Adequate organ function defined as:

   1. Creatinine < 1.6 mg/dl
   2. ALT/AST < 3x upper limit of normal range
   3. Direct bilirubin <2.0 mg/dl
   4. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea, pulse oxygen > 92% on room air, and DLCO > 40% (corrected for anemia)
   5. Left Ventricle Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO/MUGA
5. Evidence of disease by standard morphologic or by MRD criteria.
6. Male or female age ≥ 18 years.
7. ECOG Performance Status that is either 0 or 1.
8. No contraindications for leukapheresis.
9. Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria:

1. Active hepatitis B or active hepatitis C.
2. HIV Infection.
3. Class III/IV cardiovascular disability according to the New York Heart Association Classification.
4. Subjects with clinically apparent arrhythmia or arrhythmias who are not stable on medical management within two weeks of enrollment.
5. Active acute or chronic graft-versus-host disease (GVHD) requiring systemic therapy.
6. Concurrent use of systemic steroids or immunosuppressant medications. Recent or current use of inhaled steroids or physiologic replacement with hydrocortisone is not exclusionary. For additional details regarding use of steroid and immunosuppressant medications.
7. CNS3 disease that is progressive on therapy, or with CNS parenchymal lesions that might increase the risk of CNS toxicity.
8. Pregnant or nursing (lactating) women.
9. Receipt of a prior investigational study agent within 4 weeks prior to enrollment. *Note- patients who have received anti-CD19 CART cells (e.g. CART19/CTL019) on an investigational study where cell infusion occurred greater than 4 weeks before the screening visit are NOT excluded.
10. Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Frey, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Singh N, Frey NV, Engels B, Barrett DM, Shestova O, Ravikumar P, Cummins KD, Lee YG, Pajarillo R, Chun I, Shyu A, Highfill SL, Price A, Zhao L, Peng L, Granda B, Ramones M, Lu XM, Christian DA, Perazzelli J, Lacey SF, Roy NH, Burkhardt JK, Colomb F, Damra M, Abdel-Mohsen M, Liu T, Liu D, Standley DM, Young RM, Brogdon JL, Grupp SA, June CH, Maude SL, Gill S, Ruella M. Antigen-independent activation enhances the efficacy of 4-1BB-costimulated CD22 CAR T cells. Nat Med. 2021 May;27(5):842-850. doi: 10.1038/s41591-021-01326-5. Epub 2021 Apr 22. PMID 33888899